CLINICAL TRIAL: NCT07294690
Title: The Effect of Preoperative Training With Virtual Reality on Anxiety, Readiness for Surgery and Recovery Process of Patients in Colorectal Cancer Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ozkan Karadede, Nurse Practitioner, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-83045809-604.01-1017096
Record Dates: First submitted 2025-11-21; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Anxiety, Surgical Preparation, and Recovery Process in Colorectal Cancer Surgery
Keywords: colorectal surgery; Anxiety; Surgical Preparation; Recovery Process
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention)
- virtual reality group (Experimental): Patients undergoing colorectal surgery will be trained using virtual reality glasses.
  Interventions: Device: Patients undergoing colorectal surgery will be trained using virtual reality glasses.

INTERVENTIONS:
Device: Patients undergoing colorectal surgery will be trained using virtual reality glasses. — Patients undergoing colorectal surgery will be trained using virtual reality glasses.
  Arms: virtual reality group

SUMMARY:
The aim of the study is to determine the effect of The Effect of Preoperative Training with Virtual Reality on Anxiety, Readiness for Surgery and Recovery Process of Patients in Colorectal Cancer Surgery.

Research Hypotheses

In patients undergoing colorectal surgery:

H1 The comfort level of patients who received preoperative training using virtual reality is higher than that of patients who received training using written brochures and the control group.

H2. The anxiety level of patients who received preoperative education using the virtual reality method is lower than that of patients who received education via written brochures and the control group.

H3 The satisfaction level of patients who received preoperative education using the virtual reality method is lower than that of patients who received education via written brochures and the control group.

ELIGIBILITY:
Inclusion Criteria:

Agreement to participate in the study, Ability to read and write in Turkish, Being conscious and communicative.

Exclusion Criteria:

Those with any psychiatric illness, Those diagnosed with an anxiety disorder and taking medication for anxiety, Those with active nausea, vomiting, or headache, Those with vision or hearing problems, Those with a history of seizures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2025-12-09 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
(State Trait Anxiety Inventory I-II) | 24 hour
  STAI I determines how an individual feels at a specific moment and under specific conditions. The State-Trait Anxiety Inventory (STAI II) determines how individuals generally feel in their current situation and conditions.
  Inventory items are scored between 1 and 4. High scores on the inventory indicate that the person has high levels of state and trait anxiety. Scores between 0 and 19 on the inventory indicate no anxiety, 20-39 points indicate mild anxiety, 40-59 points indicate moderate anxiety, and 60-80 points indicate severe anxiety.
The Preparedness for Colorectal Cancer Surgery Questionnaire (PCSQ) | 24 hour
  The scale determines whether the verbal and written information provided about the surgery prepares individuals for the surgery. The scale is a 4-point Likert scale ranging from positive to negative. The scale consists of a total of 24 items. The score that can be obtained from the scale ranges from 0 to 96. Item 24 on the scale is reverse-scored. The scale is evaluated by calculating the total score of the items. High scores indicate a high level of readiness.
Recovery Quality-40 Survey (QoR-40) | 24 hour
  The scale consists of a total of 40 items. It comprises five subscales: emotional state, physical comfort, patient support, physical independence, and pain. The scale is a 5-point Likert scale, and items are scored on a scale of 1 to 5. Subscale averages are obtained by summing the scores for each subscale, and the total survey score is obtained by summing all items. A higher score indicates that patients' physical and emotional well-being is at the expected level (good condition) post-surgery. A low score indicates that the patient's well-being post-surgery has been negatively affected.

SECONDARY OUTCOMES:
Cortisol Level | 24 hour
  Cortisol, commonly known as the "stress hormone," is essential for life. When stress occurs, cortisol levels increase. Cortisol is secreted by the adrenal cortex in response to various stimuli. It enables the organism to adapt to its environment. Cortisol helps the organism defend against dangers by enhancing its homeostasis ability. Cortisol levels were measured using saliva samples taken at specified times.
Number of Steps | 24 hour
  A pedometer wristband was used to monitor the patient's daily physical activities and determine the number of steps taken.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data (IPD) collected in this study will be shared with other researchers for scientific purposes. The data to be shared will include anonymized demographic characteristics, outcome measures, and variables used in the analyses, with no information that could directly or indirectly identify individual participants. Data will be made available after publication of the primary study results. Access to the data will be granted upon reasonable request, subject to submission of a written scientific proposal and confirmation of compliance with ethical standards. The data will be provided through a secure external data-sharing platform, and a link to the dataset will be made available in the ClinicalTrials.gov record when accessible.